CLINICAL TRIAL: NCT02359929
Title: A Phase I Study of Mesenchymal Stromal Cells for the Treatment of Acute and Chronic Graft Versus Host Disease
Brief Title: BMT Autologous MSCs for GvHD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: CURE Foundation (Other)
Responsible Party: Principal Investigator, Muna Qayed, Assistant Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00076372
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Graft Versus Host Disease; Acute Graft Versus Host Disease; Chronic Graft Versus Host Disease
Keywords: graft versus host disease; GVHD
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1: Infusion of MSCs (Experimental): First three subjects enrolled will receive a single infusion of mesenchymal stromal cells based on their individual weight
  Interventions: Biological: Autologous mesenchymal stromal cells (MSCs)
- Dose Level 2: Infusion of MSCs (Experimental): Subsequent subjects enrolled will receive two infusions (a week apart) of mesenchymal stromal cells based on their individual weight
  Interventions: Biological: Autologous mesenchymal stromal cells (MSCs)
- Dose Level 3: Infusion of MSCs (Experimental): Subsequent subjects enrolled will receive four infusions (a week apart) of mesenchymal stromal cells based on their individual weight
  Interventions: Biological: Autologous mesenchymal stromal cells (MSCs)

INTERVENTIONS:
Biological: Autologous mesenchymal stromal cells (MSCs) — Infusion of MSCs delivered to each patient will depend on their weight and assigned dose level. The maximal individual dose of MSCs any patient will receive is 2 x 1000000 cells/kg.

SUMMARY:
Subjects in this study have had an allogeneic (blood or marrow cells from another person) blood or marrow transplant to treat leukemia, lymphoma or other cancer of the blood, and have now developed Graft Versus Host Disease (GVHD) that is not responding to standard treatment. GVHD is when the graft (transplanted bone marrow or blood) attacks the recipient's body. GVHD occurs early after transplant (acute) and/or sometimes months after transplant (chronic). Both forms can be life threatening; chronic GVHD can be a lifelong disabling condition.

Mesenchymal stromal cells (MSCs) exist in tissues throughout the body. One place they are found is in the bone marrow and from here they can be obtained by needle aspiration, the same way bone marrow samples are obtained to test for leukemia. This study uses autologous MSCs obtained from the recipient with acute and/or chronic GVHD, which have a lower chance of being rejected. These MSCs may promote tolerance, helping the donor immune cells accept the recipient's body.

This trial is being conducted as a step toward testing the long-term hypothesis that freshly cultured autologous MSC grown in platelet lysate-containing medium will modulate donor T-cell immune responses and reduce GVHD in allo-HSCT recipients. As a phase I dose escalation trial of autologous MSC in patients with acute and chronic GVHD, the main aim is to evaluate the safety of this therapy and its effects on GVHD biomarkers and T-cell phenotype

DETAILED DESCRIPTION:
EPIC MSC2014-002 solution- Autologous Mesenchymal Stromal Cells expanded using pooled human platelet lysate,is made up of autologous marrow-derived mesenchymal stromal cells ex vivo expanded numerically for approximately 14 days using pooled human Platelet Lysate (phPL), harvested from culture on the day of infusion and suspended at a concentration of 4 million cells/ml in Plasmalyte A with 0.5% human serum albumin. This is a phase I dose-escalation, open label, non-randomized, non-placebo controlled, single group assignment study to evaluate the safety and tolerability of EPIC MSC2014-002. The product will be infused intravenously and will be administered at one of three dose levels: (Dose level 1): Single Cell infusion 2 x 10^6 cells/kg, (Dose Level 2): Two weekly Cell infusions 2 x 10^6 cells/kg , (Dose level 3): Four weekly Cell infusion 2 x 10^6 cells/kg. This Phase I clinical trial will enroll 12-24 subjects with acute or chronic GVHD. The duration of this study for each patient is 1 year. The investigators anticipate that this study will be completed within 3 years of commencement.

Objectives:

* To determine the safety and tolerability of infusing escalating doses of autologous MSCs for patients with acute or chronic GVHD.
* To assess the overall response rate of acute and chronic GVHD to autologous MSC infusion. These data will be used to plan future, larger clinical trials to evaluate the efficacy of autologous MSCs for the treatment of GVHD.
* To determine the effect of MSC infusion on lymphocyte phenotype, inflammatory biomarkers and GVHD specific biomarker levels

ELIGIBILITY:
Inclusion Criteria:

* Age: patients must be ≥12 years old and weigh > (25 kg) at the time of study entry.
* Patients must have received an allogeneic stem cell transplant for a hematologic malignancy.
* Must have one of the following diagnoses:
* Acute GVHD (grade II-IV) requiring systemic therapy and refractory/unresponsive to glucocorticoid (>1 mg prednisone-equivalent/kg x 1 week)
* Chronic GVHD that is extensive and not improved despite therapy with glucocorticoid (> 0.5 mg prednisone-equivalent/kg/day) and therapeutic doses of a calcineurin inhibitor for at least 4 weeks, or worsened within 2 weeks, or overlap syndrome not responding to glucocorticoid treatment (>1 mg prednisone-equivalent/kg x 1 week)

Exclusion Criteria:

* Active invasive fungal infection requiring treatment with anti-fungal medication.
* Active viral infection requiring treatment with anti-viral medication.
* Persistence/relapse at the time of study entry of the primary malignancy for which the transplant was performed. Patients with a history of relapsed malignancy who have achieved a remission at the time of evaluation for study participation will not be excluded.
* Known T-cell donor chimerism of <50%.
* Documented DLCO <50% (if performed within 90 days of enrollment) or requirement for supplemental oxygen.
* Pregnancy or breastfeeding. Patients of childbearing capability should agree to use contraception.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of EPIC MSC2014-002 based on dose limiting toxicities (DLTs) | 6 months
  Number of adverse events that are considered dose limiting toxicities (DLTs). DLTs will be defined as any grade ≥3 adverse reaction that is unexpected, or considered attributable to the MSC infusion (attribution listed as at least probable).

SECONDARY OUTCOMES:
Overall Response Rate for acute GVHD subjects | 6 months
  Percentage of subjects that had a complete response (CR) or partial response (PR). CR is resolution of acute GVHD in all involved organs and PR is improvement of at least 1 stage without worsening in other organ systems.
Overall Response Rate for chronic GVHD subjects | 6 months
  Percentage of subjects that had a reduction in the overall National Institute of Health (NIH) score at three months, without worsening any specific organ. NIH Criteria for Clinical Trials in Chronic Graft-versus-Host Disease scale: Organs and sites to be scored include skin, mouth, eyes, gastrointestinal tract, liver, lungs, joints and fascia, and the genital tract. Each organ or site is scored according to a 4-point scale (0 to 3), with 0 representing no involvement and 3 reflecting severe impairment. Total possible score: 63
Transplant-related mortality | 6 months
  Transplant-related mortality defined as any death occurring in continuous complete remission
Incidence of Relapse | 6 months
  Percentage of subjects who experience relapse of underlying malignancy
Disease-free survival | 1 year post transplant
  Disease-free survival will be defined as survival without relapse of underlying malignancy.
Overall-survival | 1 year post transplant
  Overall-survival will be defined as survival with or without relapse of underlying malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Muna Qayed, MD, Principal Investigator — Children's Healthcare of Atlanta/Emory University
Locations (1):
- Children's Healthcare of Atlanta/Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Result] Stenger E, Giver CR, Langston A, Kota D, Das PK, Chinnadurai R, Galipeau J, Waller EK, Qayed M. Safety of autologous freshly expanded mesenchymal stromal cells for the treatment of graft-versus-host disease. Front Immunol. 2022 Sep 14;13:959658. doi: 10.3389/fimmu.2022.959658. eCollection 2022. PMID 36189324